CLINICAL TRIAL: NCT01901445
Title: Quality of Life in Children and Adolescents With Chronic Functional Constipation: Educational Action Effects
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Gabriela Cunha Schechtman Sette, PhD Student, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CAAE-0039.0.447.000-11
Record Dates: First submitted 2013-05-25; First posted 2013-07-17 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Chronic Functional Constipation
Keywords: Quality of life; Constipation; Focus groups; Health education; Problem-based learning
MeSH Terms: conditions — Constipation; Health Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational action group (Experimental)
  Interventions: Behavioral: Educational action with focal group
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Educational action with focal group
  Arms: Educational action group

SUMMARY:
The purpose of this study is to determine if the quality of life in children and adolescents diagnosed with chronic functional constipation improves after educational activity in focus group composed by these patients' mothers.

DETAILED DESCRIPTION:
The present research will be conducted on the specific constipation clinic in Hospital das Clínicas at Universidade Federal de Pernambuco.

ELIGIBILITY:
Inclusion Criteria:

* Children (6 to 9 years-old) and adolescents
* Diagnostic of chronic functional constipation

Exclusion Criteria:

* Patients using calcium and/or heme
* Patients with organic diseases that causes constipation

Ages: 6 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 11 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-08 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
The improvement in the quality of life on participants after the intervention | 3 months
  The quality of life outcomes will be assessed by using the Generic Core Questionnaires (Standard form) of Measurement Model for the Pediatric Quality of Life InventoryTM version (PedsQL) 4.0 Generic Core Scales (VARNI et al., 2001) was translated and validated in Brazil by Klatchoian et al. (2008).

SECONDARY OUTCOMES:
The improvement in clinical parameters of chronic functional constipation | 3 months
  The clinical parameters were assessed according to a specific questionnaire used on patient assistance at clinical hospital at UFPE. This questionnaire will be applied before and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Gabriela CS Sette, MSc, Principal Investigator — Universidade Federal de Pernambuco
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil